CLINICAL TRIAL: NCT07091253
Title: Objective Physical Activity and Sedentary Behaviors of People Living With HIV in New York City
Brief Title: Physical Activity and People Living With HIV in New York City
Status: Terminated | Type: Observational
Why Stopped: The PI moved to another institution. The award and program are no longer at Queens College.
Sponsor: Queens College, The City University of New York (Other)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: 62057-0050
Record Dates: First submitted 2019-08-05; First posted 2025-07-29 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV+
  Interventions: Other: HIV+

INTERVENTIONS:
Other: HIV+ — Participants living with HIV will use a triaxial accelerometer for a week in order to measure the physical activity and sedentary behaviors

SUMMARY:
The study evaluates the physical activity and sedentary behaviors, as well as the relationship between physical activity an overall health in people living with HIV (PLWH).

DETAILED DESCRIPTION:
PLWH now live longer due to the effectiveness and availability of anti-retroviral therapy (ART). However, serious physical and mental health issues are often reported in this population. Research suggests that physical activity (PA) can improve physical and mental health in PLWH. However, while studies on self-reported PA among PLWH abound, very few studies have reported on the objectively measured PA (i.e., the standard for PA assessment) and sedentary behaviors of PLWH and the relationship between PA and physical and mental health in this population. The purpose of this study are to evaluate the objectively measured PA and sedentary behaviors of PLWH in New York City, as well as the relationship between PA and overall health in this population. A better understanding of the PA and sedentary behaviors is critical to establishing PA programs that can lead to enhancement of overall health.

The study is cross-sectional in design and will last a total of one week. Participants who agree to participate will be asked to complete a series of questionnaires evaluating physical health, mental health, physical activity and nutrient intake, and will be asked to wear an accelerometer at the hip for seven consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Having an HIV diagnosis
* Able to engage in daily physical activities
* Willing to carry an accelerometer for seven days at the waist
* Living within the 5 boroughs of New York City, and
* Willing to be contacted daily by phone or text during the study.

Exclusion Criteria:

* Having an unmanaged chronic disease or musculoskeletal disease that would limit physical activity
* Having suicidal ideations
* Currently being pregnant

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People living with HIV
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Physical activity and sedentary time | one week
  Time engaged in moderate to vigorous physical activity, as well as sedentary time, during the measurement week as assessed through accelerometry.

SECONDARY OUTCOMES:
Health Status | last 30 days
  Overall health status will be assessed through 4 short questions from the Behavioral Risk Factor Surveillance System. The questions ask about the participant's perception of their current general health in a Likert scale, the number of days during the past 30 days their physical health was not good, the number of days during the past 30 days their mental health was not good and number of days in the last 30 days their physical or mental health kept them from doing their usual activities.
Exercise Vital Sign questionnaire | From enrollment to the end of the protocol at 7 days
  Self reported physical activity will be evaluated using the Exercise Vital Sign questionnaire. The questionnaire provides information on the days per week the participant engages in moderate to strenuous physical activity, and the number of minutes per day the participant engages in such behaviors. The range of days is 0 to 7, and the range of minutes per day is 0 to 1440. The number of days and the number of minutes per day that the participant engages in moderate to strenuous physical activity will be multiplied to get the total number of minutes per week that the participant engages in such activity. Less than 150 minutes per week of physical activity will be considered "not meeting physical activity guidelines for Americans", and equal or more than 150 minutes per week will be considered "meeting physical activity guidelines for Americans". The questionnaire will be administered at the beginning and at the end of the study.
Nutrient Intake Assessment | From enrollment to the end of the protocol at 7 days
  Nutrient intake will be evaluated using the Rapid Eating Assessment for Participants (REAPS) questionnaire. The questionnaire includes 16 questions. The first 13 questions are used to calculate the diet quality score. They include 3 possible answers: "usually/always"= 1 point, "sometimes"= 2 points, "rarely/never" = 3 points. The scores are added to determine diet quality on a scale of 13 (worst outcome) to 39 (best outcome). Higher scores indicating a healthier diet.
  The last 2 questions are not included in the total score calculation. One question includes "Yes" or "No" answers, and 1 question is rated on a 5-point scale ranging from 1 (best outcome) to 5 (Worst outcome).
Diagnosed Diseases | At enrollment, on the first day of the protocol.
  Participants will also be asked questions from the Behavioral Risk Factor Surveillance System about diagnosed diseases including: coronary heart disease, myocardial infarction, stroke, chronic obstructive pulmonary disease, depressive disorder and diabetes. Possible answers include: "Yes", "No", "Don't know/Not sure" or "Refused". This is done for descriptive purposes and and there is no scale or score associated with this measure.
Depressive symptoms using the Beck Depression Inventory II (BDI-II) | From enrollment to the end of the protocol at 7 days
  Depressive symptoms will be evaluated using the Beck Depression Inventory II (BDI-II). The BDI-II is a self-report questionnaire designed to assess the severity of depressive symptoms in adults and adolescents aged 13 and older during the past 2 weeks. Items are rated on a 4-point scale ranging from 0 (minimum score) to 3 (maximum score) based on severity of each item. The minimum total score is 0 and the maximum total score is 63. The higher the score the worse the severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Quiles, Ed.D., Principal Investigator — Queens College CUNY
Locations (1):
- Applied Physiology Laboratory, Flushing, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quiles NN, Balachandran A, Ortiz A. Comparison of the Exercise Vital Sign Questionnaire With Accelerometry and Physical Activity Behaviors in People Living With HIV in New York City: A Cross-Sectional Study. J Assoc Nurses AIDS Care. 2025 Dec 29. doi: 10.1097/JNC.0000000000000617. Online ahead of print. PMID 41459937